CLINICAL TRIAL: NCT01807832
Title: The Use of Capsaicin Challenge for Diagnosis, Monitoring and Follow-up of Chronic Cough.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-13-LF-0695-CTIL
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Cough
Keywords: chronic cough; cough reflex hypersensitivity; capsaicin
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chronic cough (Other): Capsaicine challenge in chronic cough patients
  Interventions: Other: capsaicin challenge

INTERVENTIONS:
Other: capsaicin challenge

SUMMARY:
The purpose of this study is to determine whether the capsaicin challenge can improve the diagnosis, treatment, monitoring and follow-up in patients with chronic cough.

DETAILED DESCRIPTION:
Capsaicin is administrated in incremental concentrations with two inhalations of normal saline solution. Patients are instructed to exhale to functional residual capacity and than to inhale through the mouthpiece for 1 second (single breath inhalation). The number of coughs in the first 10 seconds after each inhalation is counted. C2; the concentration of which the patient responded by 2 coughs, C5;the concentration of which the patient responded by 5 coughs. The challenge ends at C5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persisting cough for more than 3 months, without known respiratory or lung diseases

Exclusion Criteria:

* Diagnosis of respiratory or lung diseases of any kind

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
cough reflex hypersensitivity | 3 months